CLINICAL TRIAL: NCT01628263
Title: Does Screening Parents Allow Targeting of a Paediatric Intensive Care Follow-up Clinic? A Feasibility Study
Brief Title: Does a Follow-up Appointment Help Parents of Children on PICU?
Acronym: PICUfu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sarah Goodwin, Specialist Registrar, University Hospitals Bristol and Weston NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CH/2011/3827
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PICU; Follow up; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow up Clinic (Experimental): Participants will receive an offer of a follow up clinic two months post discharge, staffed by the unit Clinical Psychologist, a PICU doctor and PICU nurse.
  Interventions: Other: Follow up Clinic for High risk participants
- Control (No Intervention): Participants will not receive an offer of a follow up clinic

INTERVENTIONS:
Other: Follow up Clinic for High risk participants — Families where either or both parents are screened to be at risk of PTSD or depression are randomised in a 1:1 ratio to the intervention or control arm. Those in the intervention arm will receive an offer of a follow up clinic two months post discharge, staffed by the unit Clinical Psychologist, a PICU doctor and PICU nurse. Those in the control arm will not be offered a follow up clinic.
  Arms: Follow up Clinic

SUMMARY:
The aim of our study is to determine the feasibility of carrying out a randomized controlled trial (RCT) to investigate whether screening parents of children admitted to pediatric intensive care unit (PICU) so as to target follow-up at those most at risk of developing posttraumatic stress disorder (PTSD), is effective at reducing adverse psychological sequelae.

DETAILED DESCRIPTION:
The study will assess the feasibility of offering a follow up clinic to parents identified to be vulnerable for future psychological difficulties after their child's admission to the Paediatric Intensive Care Unit (PICU) at Bristol Children's Hospital. Both mothers and fathers of children admitted to PICY for a duration of at least 12 hours will be invited to participate in this study. Screening measures will be used to identify vulnerability to future post-traumatic stress disorder (PTSD) and depression. Where one or both of the parents has been scored as high risk they will be randomised to receive the intervention or the control arm of the study (ratio 1:1). The intervention involves a follow-up clinic two months pots admission, staffed by the unit Clinical Psychologist, a PICU doctor and PICU nurse. In the control arm no follow-up clinic will be offered (i.e. current standard care).

Objectives:

i) To investigate the recruitment rates, clinic attendance and follow-up rates in order to perform an accurate sample size calculation for a larger study.

ii) To carry out initial statistical analysis to estimate the odds ratio and 95% confidence interval of developing PTSD, anxiety and depression after being offered the follow-up intervention as opposed to not being offered it.

iii) To assess the acceptability of providing targeted follow-up both to those who receive it and those who are excluded due to low risk.

The study is of importance to the public because not only does PTSD negatively affect quality of life, it is also associated with increased use of health care services and resources.

ELIGIBILITY:
Inclusion Criteria:

* All parents of children admitted to paediatric intensive care for over 12 hours.

Exclusion Criteria:

* Parents deemed unsuitable for the study by the responsible consultant. This will include families where a child's condition is suspected to result from non-accidental injury or where withdrawal of care is being discussed due to a child's critical condition. Families will be excluded if their child died during or after admission, as these families are already followed up routinely.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The Impact of Event Scale-Revised (IES-R) | 5 months post discharge
  Widely used self-report measure of responses to trauma
Hospital Anxiety & Depression Scale (HADS) | 5 months post discharge
  Widely used self-report measure of anxiety and depression

SECONDARY OUTCOMES:
Feedback Questionnaire | 6 months post discharge
  Questionnaire to elicit feelings about taking part in the study including questions about acceptability of completing screening measures and some people being excluded from clinic due to being low risk. Clinic attenders will be asked if they found it a useful experience and how it could be improved.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Goodwin, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust; Victoria Samuel, Study Director — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (1):
- Bristol Royal Hospital for Children, Bristol, United Kingdom